CLINICAL TRIAL: NCT07396025
Title: Evaluation of the Effectiveness of Surgical and Diagnostic Techniques in Patients With Steno-occlusive Diseases of the Cerebral Vessels
Brief Title: Effectiveness of Surgical and Diagnostic Methods in Cerebral Vascular Occlusive Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Centre for Neurosurgery, Republic of Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26100905; AP26100905 (Other Grant/Funding Number: Science Committee of the Ministry of Science and higher education of the Republic of Kazakhstan)
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carotid Artery Occlusion
Keywords: stroke, carotid artery occlusion, cerebral bypass, STA-MCA bypass, atherosclerosis, CT and MRI perfusion, cerebral angiography; stroke; carotid artery occlusion; cerebral bypass; STA-MCA bypass; atherosclerosis; CT and MRI perfusion; cerebral angiograph
MeSH Terms: conditions — Stroke; Atherosclerosis | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with chronic occlusive internal carotid artery cerebrovascular disease (Other)
  Interventions: Procedure: Revascularization/Conservative management

INTERVENTIONS:
Procedure: Revascularization/Conservative management — This study attempts to improve surgical treatment outcomes among people with chronic carotid artery occlusive disease by conducting a comprehensive review of neuroradiological, clinical, and cognitive data. The evaluation involves an extensive angiographic analysis, including pre- and postoperative measurements of superficial temporal artery branch diameters, assessment of the Circle of Willis and collateral pathways, alongside cerebral perfusion metrics, cognitive status, and clinical outcomes. Major focus is directed towards evaluating the degree of intracranial revascularization following to extracranial-intracranial bypass by postoperative angiographic evaluations.

SUMMARY:
This study attempts to improve surgical treatment outcomes among people with chronic carotid artery occlusive disease by conducting a comprehensive review of neuroradiological, clinical, and cognitive data. The evaluation involves an extensive angiographic analysis, including pre- and postoperative measurements of superficial temporal artery branch diameters, assessment of the Circle of Willis and collateral pathways, alongside cerebral perfusion metrics, cognitive status, and clinical outcomes. Major focus is directed towards evaluating the degree of intracranial revascularization following to extracranial-intracranial bypass by postoperative angiographic evaluations. This integrative strategy aims to refine surgical reasons, better predictions of functional and cognitive outcomes, minimize postoperative risks, and eventually improve the overall efficacy of treatment in this patient population.

DETAILED DESCRIPTION:
Patient selection. Patients with asymptomatic or symptomatic ICA occlusion undergoing STA-MCA bypass at the neurosurgical center will be prospectively enrolled between August 2025 and December 2027. Prior to registration, all participants will provide written informed permission in compliance of the Declaration of Helsinki's ethical guidelines.

Preoperative evaluation will include computed tomography angiography (CTA), magnetic resonance imaging (MRI), digital subtraction angiography (DSA), and comprehensive neurological and neuropsychological assessments. Magnetic Resonance Imaging also will be employed to exclude patients with extensive territorial infarctions. Only patients with radiologically confirmed ICA occlusion and arterial spin labeling (ASL) MRI-documented cerebral hypoperfusion in the affected vascular territory who undergo STA-MCA bypass will be included.

The study cohort will be recruited at the National Center for Neurosurgery in Astana through a multidisciplinary collaboration involving neurosurgeons, radiologists, neurologists, and neuropsychologists. All data will be collected using standardized case report forms and subsequently entered into a unified, secure database. Patient confidentiality will be ensured through strict coding and anonymization of personal identifiers and medical record identification numbers (MRINs).

Study variables. Data collection will include the following variables:

Demographic characteristics: Age, gender, birthplace, nationality, employment status, profession, and education level. Medical history: Past medical and surgical history, onset of TIA or stroke, vascular risk factors (hypertension, diabetes mellitus, dyslipidemia, atrial fibrillation), comorbidities (including genetic disorders), previous surgeries, ongoing follow-up care, current medications, and BMI. Clinical, neurological, and cognitive status: Baseline neurological examination findings, Modified Rankin Scale (mRS) and National Institutes of Health Stroke Scale (NIHSS) scores, history of seizures, quality-of-life measures, cognitive reserve indicators (educational attainment and occupational complexity), and engagement in cognitively stimulating activities will be assessed. Lifestyle factors: Smoking status, dietary habits, physical activity, alcohol consumption, sleep quality, vacation frequency, tobacco use, and other lifestyle factors. Radiological and hemodynamic parameters: Location and length of the internal carotid artery occlusion; collateral circulation patterns; Circle of Willis configuration; ASL perfusion metrics; cerebral blood flow (CBF) asymmetry indices; infarct burden; white matter hyperintensities; and postoperative bypass patency and the diameter of STA pre and postoperatively.

Study procedures. To evaluate the ICA occlusion, a three-level assessment will be conducted using instrumental methods. This comprehensive approach includes CTA of the head and neck vessels, specialized MRI ASL and Time-of-flight (TOF) sequences, and a confirmatory assessment of occlusion during DSA. All imaging studies will be performed and interpreted by experienced neuroradiologists and neurosurgeons, with findings reviewed collaboratively.

All patients will undergo CTA of the head and neck vessels with a slice thickness of 0.5-0.625 mm to confirm internal carotid artery occlusion and to measure the diameter of the donor STA branch at 2 mm distal to its bifurcation.

To evaluate cerebral blood flow (CBF) and determine the extent of cerebrovascular insufficiency, MRI perfusion studies will be conducted before surgery on 1,5 or 3 Tesla MRI. The main perfusion method will be ASL, which will provide quantitative CBF values, assess the degree of perfusion deficit, and reveal signs of compensatory collateral circulation based on the presence of arterial transit artifacts (ATA). Selective cerebral angiography will be performed using a biplane digital subtraction angiography system (Artis Zee, Siemens) with a 6F guiding catheter at a frame rate of 7.5 frames per second. The angiographic assessment will evaluate the presence of communicating arteries, the completeness of the Circle of Willis, and the extent of collateral circulation. Hemodynamic compensation will be quantified by analyzing filling times and phase delays across the arterial, parenchymal, and venous phases, expressed in frames. Image analysis will be conducted using Siemens Artis Q angiography software to ensure accurate and reproducible measurements.

Neurological status assessment. The degree of neurological deficit before and after surgery will be evaluated by neurologist using the Baseline neurological examination findings, Modified Rankin Scale (mRS) and National Institutes of Health Stroke Scale (NIHSS) scores). The consequences of prior stroke will also be assessed with the modified Rankin Scale (mRS)15 and the Functional Activities Questionnaire (FAQ)16. Preoperatively and six months after surgery, all patients will be evaluated under a unified diagnostic protocol, with results collected and recorded separately before entering them into a general database with strict personal data encoding.

Cognitive function assessment. Changes in cognitive function before and after surgery and six months postoperatively will be assessed using the neuropsychological tests, measuring both verbal and non-verbal IQ. A standardized battery of neuropsychological tests will be administered by a psychologist to evaluate global cognition, memory, visuospatial skills, and executive function. The Montreal Cognitive Assessment (MoCA) will be used as a screening tool for global cognitive function, assessing domains including attention, executive functions, memory, language, visuospatial skills, abstraction, and orientation17. The Rey Auditory Verbal Learning Test (RAVLT) will be employed to evaluate verbal learning and memory performance, including immediate recall, delayed recall, and recognition memory18. Nonverbal test of Kohs Block Design will be used to assess visuospatial reasoning, problem-solving, and perceptual-motor coordination by requiring participants to reproduce geometric patterns with colored blocks19. The Stroop Test will be applied to measure selective attention, processing speed, and cognitive flexibility by evaluating the ability to inhibit cognitive interference20.

Treatment. All eligible patients with ICA occlusion will undergo standard STA-MCA bypass surgery performed by experienced neurosurgeons. The procedure will be carried out using a standardized microsurgical end-to-side anastomosis technique, which is well established and routinely performed by the participating surgeons21. Intraoperative selection of the donor STA branch and recipient MCA segment will be based on vessel diameter, flow characteristics, and surgical accessibility. Intraoperative bypass patency will be assessed using the "faucet" technique21 in combination with microscopic indocyanine green (ICG) angiography to ensure adequate flow through the anastomosis.

Intraoperative perfusion and blood flow direction assessment Intraoperative perfusion and blood flow direction will be assessed using indocyanine green fluorescent angiography with the Karl Zeiss Pentera 8000 microscope equipped with FLOW 800 technology, which allows real-time visualization of cerebral vessels. All data will be processed and analyzed to create a color map depicting hemodynamic and perfusion delays. This enables comparison of perfusion parameters in the anastomosis region before and after bypass surgery, as well as assessment of blood flow direction and hyperperfusion zones in the brain. The assessment will be performed by neurosurgeons.

Postoperative study procedures.Within 1-3 days after surgery, CTA of the head and neck will be performed to confirm bypass patency, measure the caliber of the donor STA branch, and visualize its course. At 3-5 days postoperatively, ASL-based MR perfusion imaging will be conducted to evaluate cerebral perfusion changes compared with preoperative studies. 3D segmentation and quantitative perfusion mapping will be applied to provide objective assessment of regional perfusion improvements following surgery. Prior to hospital discharge, all patients will undergo a repeat evaluation of neurological status and cognitive function using the same standardized tests as preoperatively.

Follow-up assessment. At six months after surgery, all patients will undergo follow-up assessment including CTA of the head and neck to evaluate bypass patency and measure the caliber of the donor STA branch, MR perfusion imaging with 3D segmentation to assess cerebral perfusion changes, and repeat neurological and neuropsychological evaluations using the same tests administered preoperatively and at discharge (NIHSS, mRS, MoCA, RAVLT, Kohs Block Design, and Stroop tests).

Endpoint evaluation

Primary endpoints (early postoperative assessment):

1. Bypass patency assessed by CTA within 1-3 days postoperatively.
2. Cerebral perfusion improvement evaluated by ASL MR perfusion imaging 3-5 days postoperatively, including 3D segmentation and quantitative perfusion mapping, as well as assessment for the presence of cerebral hyperperfusion syndrome.
3. Surgical safety outcomes, including perioperative stroke, transient ischemic attack (TIA), or other procedure-related complications.

Secondary endpoints (six-month follow-up):

1. Clinical outcomes: Occurrence of any stroke events or death.
2. Imaging outcomes: CTA of the head and neck to assess long-term bypass patency and measure the caliber of the donor STA branch and MR perfusion imaging wit to evaluate sustained cerebral perfusion changes.
3. Functional and cognitive function improvements: Neurological and neuropsychological assessments using the same standardized tests as preoperatively and at discharge.
4. MRI perfusions pre and postoperatively after 6 months will be compared in 3 D program models and correlated with neurological and cognitive changes, and additional correlations with donor branch of STA Data processing. All collected data will be meticulously entered into a database, where revascularization progress, the development of collateral circulation, and perfusion changes correlated with neurological and cognitive shifts will be evaluated. All data will undergo statistical processing and analysis to identify patterns and correlations, as well as survival analysis to assess collateral development and psychoneurological dynamics. All participants are expected to complete study visits over the planned 6-months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ICA occlusion confirmed by CTA, MRA, and cerebral DSA.
2. MRI ASL-confirmed hypoperfusion in the territory of the occluded ICA (decrease of ≥30% compared with the contralateral side)
3. Language comprehension is preserved, with mild or no motor aphasia and no significant cognitive impairment.
4. Patients aged from 18 to 80 years.
5. Modified Rankin Scale (mRS) score 0-2.
6. Informed consent is available from the patient or legal guardian.
7. Accessible and reliable patients for follow-up

Exclusion Criteria:

1. Patients with large territorial infarction or marked cerebral atrophy on MRI.
2. No evidence of regional hypoperfusion on ASL MRI relative to the contralateral hemisphere.
3. Patients with a non-functioning STA-MCA bypass
4. Patients aged under 18
5. Patients with severe somatic conditions or mRS score > 3
6. Patients with bilateral ICA occlusion, neurovascular disease (cerebral aneurysm or arteriovenous malformation)
7. Patients with Contraindications to MRI, CTA, or DSA
8. Cardiac conditions associated with a high risk of cerebral embolism, including prosthetic heart valves, infective endocarditis, intracardiac thrombus, sick sinus syndrome, cardiac myxoma, or cardiomyopathy with left ventricular ejection fraction <25% (atrial fibrillation, patent foramen ovale, and atrial septal aneurysm are not exclusion criteria).
9. Severe systemic comorbidities, life expectancy <2 years, or a modified Rankin Scale (mRS) score >3.
10. Pregnancy.
11. Contraindications to MRI, CTA, DSA, iodinated contrast agents, or antiplatelet therapy required in the perioperative period.
12. Participation in another interventional or experimental trial within the previous 12 months, including studies involving ionizing radiation

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
STA-MCA bypass patency | From enrollment to the further follow-up of 6, 12, and 24 months.
  Patency of the extracranial-intracranial bypass will be assessed using CTA of the head and neck and classified as patent or occluded.
Donor superficial temporal artery caliber | 6, 12, and 24 months after surgery
  Diameter of the donor superficial temporal artery branch at the anastomosis site measured using CTA imaging.
Cerebral perfusion changes | 6, 12, and 24 months after surgery
  Quantitative cerebral perfusion parameters assessed using MR perfusion imaging with 3D segmentation and compared with preoperative baseline values.

SECONDARY OUTCOMES:
Global cognitive function | Preoperatively; at discharge; 6, 12, and 24 months after surgery
  Cognitive performance assessed using the Montreal Cognitive Assessment (MoCA).

OTHER OUTCOMES:
Verbal memory performance | Preoperatively; at discharge; 6, 12, and 24 months after surgery
  Verbal learning and memory assessed using the Rey Auditory Verbal Learning Test (RAVLT).
Visuospatial and executive function | Preoperatively; at discharge; 6, 12, and 24 months after surgery
  Visuospatial and executive function assessed using the Kohs Block Design Test.
Cognitive control and processing speed | Preoperatively; at discharge; 6, 12, and 24 months after surgery
  Cognitive control and processing speed assessed using the Stroop Color-Word Test.

CONTACTS AND LOCATIONS:
Locations (1):
- National Centre for Neurosurgery, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided